CLINICAL TRIAL: NCT06820346
Title: New Manual Test for the Assessment of Hip Abductor Extensibility: a Pilot Study on Precision and Accuracy
Brief Title: New Manual Test for Hip Abductor Extensibility
Acronym: 2MOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manusapiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2MOT
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy adults (Experimental): Manual and instrumental evaluation of hip adduction
  Interventions: Other: Manual and instrumental evaluation of hip adduction

INTERVENTIONS:
Other: Manual and instrumental evaluation of hip adduction — The intervention consists of a new manual test for assessing iliotibial band (ITB) tension and hip abductor extensibility. The patient lies supine on the edge of a treatment table with the non-tested leg flexed at the hip and knee, stabilizing the pelvis. The tested leg remains extended. The examiner stabilizes the non-tested leg with one hand and adducts the tested leg until a resistance is felt, ensuring no pain. The hip adduction angle is visually assessed and recorded. A subset of participants also undergoes the modified Ober test for comparison. Inertial motion sensors are used to validate the accuracy of visual assessments. The primary outcomes include intra-rater and inter-rater reliability, while secondary outcomes evaluate the test's accuracy and pelvic movement reduction.

SUMMARY:
This pilot study aims to evaluate the precision and accuracy of a new manual test for assessing hip abductor extensibility. The iliotibial band (ITB) and hip abductor muscles play a crucial role in lower limb biomechanics, and their flexibility is commonly assessed using the Ober test. However, the Ober test has limitations, including excessive pelvic movement and reliance on qualitative evaluation. This study introduces and validates a novel manual test designed to improve the accuracy and reliability of hip abductor extensibility assessment.

The primary objective is to determine the intra-rater and inter-rater reliability of the new test, measured using the intraclass correlation coefficient (ICC). The secondary objective is to compare the test's accuracy against an inertial motion sensor system and to quantify pelvic movement during the new test. To provide a comparative measure of pelvic motion, a subgroup of participants will also undergo the modified Ober test.

Forty healthy participants (20 males and 20 females) aged 18 to 30 years will be recruited. Each participant will undergo the new test, performed by two independent raters. A subset of participants will also be evaluated using the modified Ober test to assess differences in pelvic movement. Inertial sensors will be used to measure hip adduction angles and pelvic motion. Statistical analyses will include ICC calculations for reliability and paired t-tests to compare pelvic movement between the tests.

This study aims to establish a more precise and objective method for evaluating hip abductor extensibility, which may enhance clinical assessment and management of conditions associated with iliotibial band tension.

DETAILED DESCRIPTION:
This study aims to evaluate the reliability and accuracy of a new manual test for assessing iliotibial band (ITB) tension. The current standard for ITB extensibility assessment, the modified Ober test, presents limitations such as excessive pelvic movement and qualitative evaluation. The newly proposed test seeks to address these issues by minimizing extraneous movement and providing a more controlled and reproducible measurement of hip adduction.

Study Design The study follows a repeated-measures design, where intra-rater and inter-rater reliability are the primary outcomes, measured using the intraclass correlation coefficient (ICC). Secondary outcomes include the accuracy of the new test compared to an inertial motion sensor and an analysis of pelvic movement during the new test versus the modified Ober test in a subset of participants.

Participants A total of 40 healthy adults (20 males and 20 females), aged between 18 and 30 years, were recruited. The only exclusion criterion was the presence of symptomatic lower limb conditions that could interfere with the measurement, such as ligament injuries or degenerative joint diseases. No additional selection criteria were imposed, as existing literature does not categorize ITB extensibility based on age, sex, or pathology.

New Test Execution

The new test was originally proposed by Colonna (2012) and is designed to provide a more reliable and precise measurement of ITB tension. The test procedure consists of the following steps:

* Patient Positioning: The patient lies supine on the edge of a treatment table, with the non-tested leg flexed at the hip and knee, stabilizing the pelvis by resting the lateral malleolus against the table edge. The tested leg remains extended.
* Operator Positioning: The operator stands on the opposite side of the tested leg, stabilizing the knee of the non-tested leg with one hand and grasping the ankle of the tested leg with the other.
* Hip Adduction: The tested leg is gently adducted until a determined resistance is felt or the patient reports discomfort, ensuring no pain occurs.
* Measurement: The hip adduction angle is visually assessed and assigned a degree value.

This procedure is designed to enhance measurement accuracy by providing a clear and stable reference point while reducing the risk of excessive pelvic movement.

Modified Ober Test Execution A subset of participants underwent the modified Ober test for comparison. The patient lay on the side with the lower leg flexed at the hip and knee, while the upper leg remained extended. The therapist stabilized the pelvis while abducting and extending the hip, then allowing passive adduction. A goniometer was used to obtain quantitative measurements of hip adduction angles. The modified Ober test was chosen over the classic Ober test as it reduces the influence of knee flexors and patellar tension, providing a more specific assessment of ITB extensibility.

Phases of the Study

The study was conducted in six phases:

* Agreement on Measurement Methodology: Standardization of the new test and the modified Ober test procedures.
* Recruitment: Participants were enrolled at the OSCE (Osteopathic Spine Center Education) school of osteopathy in Bologna, Italy.
* Training Phase: Operators practiced test execution using a goniometer and dynamometer (100N force standardization), validated their visual assessments with inertial sensors, and refined their technique.
* Preliminary Testing for Agreement: Ten participants underwent preliminary tests to confirm measurement consistency.
* Official Data Collection: Each operator conducted the new test on both lower limbs of each participant at two time points (T0 and T1), with a minimum four-hour interval. The modified Ober test was performed on 20 participants by one operator for pelvic movement comparison.
* Data Analysis: Reliability and accuracy of the new test were assessed by comparing results to the modified Ober test and inertial sensor data.

Measurement Instruments

- Hip adduction angles and pelvic rotation were measured using Xsens® inertial sensors. These wireless sensors, placed on the pelvis and thigh, provided real-time kinematic data to validate the accuracy of visual assessments and quantify pelvic movement.

Statistical Analysis

Data were analyzed using SPSS software. Reliability was assessed using ICC values, interpreted as follows:

Below 0.5: Poor reliability 0.5 to 0.75: Moderate reliability 0.75 to 0.9: Good reliability Above 0.9: Excellent reliability Accuracy of the new test was determined by comparing operator assessments with inertial sensor data. Paired t-tests were used to compare pelvic movement between the new test and the modified Ober test, with statistical significance set at p < 0.05.

By addressing the limitations of the modified Ober test, this study seeks to introduce a more precise and clinically applicable method for assessing ITB extensibility.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects

Exclusion Criteria:

* absence of symptomatic lower limb conditions that could impede measurement, such as ligament injuries of the knee or degenerative joint diseases of the hip

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Precison of visual hip adduction evaluation | 15 seconds for each evaluation (day 1)
  intra-day concordance intra and inter examiners of the visual identification of the degrees of hip adduction by means of intraclass correlation coefficient
Accuracy of visual hip adduction evaluation | 15 seconds for each evaluation (day 1)
  Concordance intra-day between the visual and instrumental evaluation of the degrees of hip adduction. The instrumental data are obtained using a Xsens inertial sensors, which measure hip adduction angles. The sensor is placed on the shank of the tested leg, providing objective kinematic data. The concordance between the two methods is evaluated with the intraclass correlation coefficient.

SECONDARY OUTCOMES:
Pelvis rotation during hip adduction evaluation | 15 seconds for each evaluation (day 1)
  Degrees of pelvis rotation during hip adduction evaluation measured with Xsens inertial sensors, both during the new test and the modified Ober test. The average values will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Spine Center, Bologna, Bologna, Italy